CLINICAL TRIAL: NCT05784376
Title: The Southern Italian Children, Adolescents and PaRents COhort Study on Nutrition and Health
Acronym: ICARO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Collaborators: Universita degli Studi di Catania (Other)
Responsible Party: Principal Investigator, Marialaura Bonaccio, Principal Investigator, Neuromed IRCCS
Other Study IDs: DEP_012023
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Diet Habit; Diet, Healthy; Child Obesity; Parents; Nutrition, Healthy
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Education-based — Nutrition education delivered via text messages through mobile applications (e.g. WhatsApp).

SUMMARY:
Childhood obesity is a major public health concern worldwide and parents play a powerful role in children's eating behaviour. Most prior studies analysed parents and children's diet almost exclusively by evaluating food composition (i.e. calorie, macro- and micronutrient contents), with no or little attention paid to degree of food processing. The NOVA classification was proposed as a novel way to look at foods based on the degree of processing of foods rather than on their nutritional composition, postulating that processing may be as relevant to health as food composition. The term ultra-processed food (UPF) indicates industrially manufactured ready-to-eat or ready-to-heat formulations made mostly or entirely from substances extracted from foods or derived from food constituents often containing added flavours, colours, emulsifiers and other cosmetic additives. Most importantly, these industrial formulations are designed to maximize palatability and consumption through a combination of calorie-dense ingredients and chemical additives. Robust and well-conducted cohort studies worldwide found that a large dietary share of UPF is associated with shorter survival and an increased risk of non-communicable diseases. Given the rising popularity of UPF globally, and also in Mediterranean countries, the issue of food processing should be prioritized in relevant dietary recommendations with emphasis on consumption of minimally/unprocessed foods.

DETAILED DESCRIPTION:
Childhood obesity is a major public health concern worldwide and parents play a powerful role in children's eating behaviour. Most prior studies analysed parents and children's diet almost exclusively by evaluating food composition (i.e. calorie, macro- and micronutrient contents), with no or little attention paid to degree of food processing. The NOVA classification was proposed as a novel way to look at foods based on the degree of processing of foods rather than on their nutritional composition, postulating that processing may be as relevant to health as food composition. The term ultra-processed food (UPF) indicates industrially manufactured ready-to-eat or ready-to-heat formulations made mostly or entirely from substances extracted from foods or derived from food constituents often containing added flavours, colours, emulsifiers and other cosmetic additives. Most importantly, these industrial formulations are designed to maximize palatability and consumption through a combination of calorie-dense ingredients and chemical additives. Robust and well-conducted cohort studies worldwide found that a large dietary share of UPF is associated with shorter survival and an increased risk of non-communicable diseases. Given the rising popularity of UPF globally, and also in Mediterranean countries, the issue of food processing should be prioritized in relevant dietary recommendations with emphasis on consumption of minimally/unprocessed foods.

The ICARO study consists of two parts, namely Study 1 (observational) and Study 2 (intervention Study).

The main objectives of the ICARO Study (Study 1) are to:

1. Evaluate the diet of participants (i.e. children, adolescents and their parents/caregivers) in terms of food composition (i.e. calorie, macro- and micronutrient contents) and complemented by a timely and innovative approach based on the evaluation of food processing, in line with the notion that the nutrient balance of a food is only a small part of its overall health potential (10);
2. Investigate major demographic, socioeconomic, behavioural, psychosocial, and other environmental factors as potential correlates of diet and diet-related habits of both children, adolescents and parents;
3. Analyse parental influence (e.g. food attitudes and knowledge) on children and adolescents diet quality and eating habits.

Within the ICARO Study population, an Intervention Study (Study 2) is planned to increase awareness and promote adherence to a minimally-processed Mediterranean Diet and reduce the dietary share of UPFs at family level.

ELIGIBILITY:
Inclusion Criteria:

* parents/caregivers of 2-13 years old children, and adolescents aged 14-18 years at recruitment residing in Southern Italy.

Exclusion Criteria:

* not being fluent in Italian language;
* refusal to sign informed consent;
* lack of an electronic device with internet access (i.e. computer, mobile phone).

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The Southern Italian Children, Adolescents and PaRents COhort Study on Nutrition and Health (ICARO Study) is designed as a web-based prospective cohort of children, adolescents and their parents/caregivers residing in Southern Italy. Participants' data will be collected through on-line questionnaires available on the Study's website, and updated every 6 months (i.e. dietary intake, anthropometric data and health status) or yearly (i.e. socio-demographics, lifestyle, and other environmental factors). Participants will be recruited through multimedia campaigns (regional newspapers, internet, social networks), contacts with schools also through the regional school system, professional channels (e.g. paediatricians, general practitioners), and targeted meetings with the general population.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Consumption of UPF in both parents and kids (changes in) | 6 months
  3-day food records
Nutrition knowledge levels of parents (changes in) | 6 months
  Questionnaire to evaluate nutrition knowledge of parents
Body weight of both parent and kids (>14 years) (changes in) | 6 months
  self-reported height and weight

SECONDARY OUTCOMES:
Adherence to the Mediterranean Diet in both parents and kids (changes in) | 6 months
  Mediterranean Diet Screener and data from 3-day food records
Parental feeding practices (changes in) | 6 months
  Questionnaire to evaluate parental feeding practices
Psychological distress in parents (changes in) | 6 months
  12-Item General Health Questionnaire (GHQ-12)

CONTACTS AND LOCATIONS:
Overall Officials: Marialaura Bonaccio, PhD, Principal Investigator — IRCCS Istituto Neurologico Mediterraneo Neuromed; Licia Iacoviello, MD, PhD, Principal Investigator — IRCCS Istituto Neurologico Mediterraneo Neuromed

IPD SHARING:
Plan to Share IPD: Undecided